CLINICAL TRIAL: NCT03490071
Title: Three and Seven Year Follow-up of Patients Reported Symptoms, Function and Quality of Life in Patients With Longstanding Hip and Groin Pain Referred to Tertiary Care. A Longitudinal Study
Brief Title: Long-term Follow up of Patients With Longstanding Hip and Groin Pain
Acronym: Lund LHGP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lund University (Other)
Responsible Party: Sponsor
Other Study IDs: Lund LHGP
Record Dates: First submitted 2018-03-28; First posted 2018-04-06 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Hip Pain Chronic
Keywords: Longstanding hip and groin pain; Patient reported outcome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this longitudinal cohort study including young to middle aged people with longstanding hip and groin pain (LHGP) referred to tertiary care, we will collect data of patient reported symptoms, function and quality of life three and seven years after the initial contact with orthopedic surgeon.

DETAILED DESCRIPTION:
81 physically active patients (18-55 years) with (LHGP) who were enrolled in a cross-sectional study (Diagnosis and functional limitations in the young to middle-aged physically active population with long-standing hip/groin pain: A cross-sectional study) during the period October 2014 to January 2017 will be recruited to this longitudinal cohort study.

A research coordinator will contact the patients and provide them with written and oral information about the study. Patients who accept to participate will electronically complete the following questionnaires. The same questionnaires were included at baseline, i.e., in the cross-sectional study.

* Copenhagen Hip and Groin Outcome Score (HAGOS)
* HSAS - Hip Sports Activity Scale (HSAS)
* Patient Specific Functional Scale
* Medical Outcomes Study short form 36 (SF-36)
* K-10 questionnaire
* Self-Presentation in Exercise Questionnaire (SPEQ)
* Multidimensional Scale of Perceived Social Support (MSPSS)

Additional questions about treatment, medication, patient satisfaction and perceived change in hip function will be included.

For descriptive purposes, the mean difference (95% CI), or median (quartiles), between baseline and follow-up assessments will be used as appropriate. Separate linear regression models will be used to evaluate the change in each variable compared to baseline values.

ELIGIBILITY:
At baseline, the following inclusion and exclusion criteria were used:

Inclusion criteria:

* Unilateral or bilateral hip/groin pain >3 months
* Age 18-55 years
* No previous hip surgery

Exclusion criteria:

* Hip pathology (i.e., Perthes' disease)
* Verified moderate or severe osteoarthritis (OA) (Tönnis grade >1)
* Palpable hernia
* Low-back pain with a positive Lasègue test
* MRI-verified lower back/spine pathology (i.e., spinal stenosis, disc herniation)
* Other musculoskeletal co-morbidities overriding the hip-related symptoms and dysfunction
* Co-morbidities excluding physical activity and training
* Psycho-social disorders
* Drug abuse
* Not understanding the language of interest.

Ages: 18 Years to 55 Years | Sex: All
Age Groups: Adult
Study Population: Patients will be recruited from the Department of Orthopedics, Skåne University Hospital, Sweden.
Sampling Method: Non-Probability Sample
Enrollment: 81 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in the Copenhagen Hip and Groin Outcome Score (HAGOS) | 3 and 7 years after baseline (cross-sectional study)
  Patient reported outcome regarding hip dysfunction, which includes six subscales; pain, symptoms, physical function in daily living, physical function in sport and recreation, participation in physical activity, and quality of life. The score for each subscale ranges from 0-100, where 0 indicates extreme problems and 100 no problems. Patient Acceptable Symptom State (PASS) will be derived from HAGOS score using previously described cut-off values for the different subscales

SECONDARY OUTCOMES:
HSAS - Hip Sports Activity Scale (HSAS) | 3 and 7 years after baseline (cross-sectional study)
  Patient reported outcome regarding activity level. The scale ranges från 0-8 where 0 indicates the lowest activity and 8 the highest.
K-10 questionnaire | 3 years after baseline (cross-sectional study)
  Patient reported outcome regarding mental health. This instrument consists of 10 questions, where each question is scored from 1 to 5. The total score is summerized and ranges from 10 to 50, where 10 indicates no problem and 50 severe problems.
Self-Presentation in Exercise Questionnaire (SPEQ) | 3 years after baseline (cross-sectional study)
  Patient reported outcome regarding self image during exercise and consists of 14 questions. Each question is assessed on a 6-point Likert-type scale ranging from 1 (strongly disagree) to 6 (strongly agree). Higher scores represent a greater desire to present oneself as an exerciser and a greater use of strategies to portray oneself as an exerciser.
The Multidimensional Scale of Perceived Social Support (MSPSS) | 3 years after baseline (cross-sectional study)
  The Multidimensional Scale of Perceived Social Support (MSPSS) is designed to measure perceptions of support from 3 sources: Family, Friends, and a Significant Other. The scale is comprised of a total of 12 items, with 4 items for each subscale. The items are scored on 7 point likert scale anging from 1 (very strongly disagree) to 7 (very strongly agree). The mean value tor each subscale are calculated. High score indicates a percetion of good social support.
Medical Outcomes Study short form 36 (SF-36) | 3 and 7 years after baseline (cross-sectional study)
  Patient reported outcome regarding general health, which includes eight subscales; vitality, physical functioning, bodily pain, general health perception, physical role functioning, emotional role functioning, social role functioning and mental health. The score for each subscale ranges from 0-100, where 0 indicates extreme problems and 100 no problems.
Additional questions regarding treatment, medication, patient satisfaction and perceived change in hip function. | 3 and 7 years after baseline (cross-sectional study)
  Additional questions about treatment, medication, patient satisfaction and perceived change in hip function will be included for descriptive purpose.

OTHER OUTCOMES:
Imaging | 7 years after baseline
  Plain radiographs with an anterior-posterior projection and Dunn-projection to evaluate hip morphology and detect possible signs of osteoarthrosis.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Ageberg, PhD, Principal Investigator — Lund University
Locations (1):
- Department of Health Sciences, Lund University, Lund, Sweden

IPD SHARING:
Plan to Share IPD: Undecided